CLINICAL TRIAL: NCT06563466
Title: PEGASUS - Improving Treatment for Patients with Emotionally Unstable Personality Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Principal Investigator, Carsten Hjorthøj, Associate Professor, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEGASUS EUPD; 3166-00026B (Other Grant/Funding Number: Independent Research Fund Denmark)
Record Dates: First submitted 2024-08-19; First posted 2024-08-20 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Borderline Personality Disorder; Relatives
Keywords: Borderline Personality Disorder; Relatives; Group psychotherapy; Case management; Psychoeducation; Family; Caregiver
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Case Managers; Therapeutics

STUDY DESIGN:
Intervention Model Description: We have planned a single blinded randomized controlled trial (RCT) pilot study. The group of participating patients and their participating relatives will be randomized into treatment as usual (TAU) or to receive the additional PEGASUS intervention, and we will be comparing the two groups. The randomization will be made 1:1 and created in the randomization module in REDCap with a block-size unknown to the assessors. Since we are conducting a pilot study, sample size is small, and we won't be able to create a stratified randomization.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators, outcome assessor and statistician will be blinded. Because of the nature of this study, it will not be possible to blind the participant or therapists providing the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment as usual (TAU) (Active Comparator): Patients with BPD are offered group-based treatment and individual therapy according to the standardized healthcare delivery models, known as the "psychiatric treatment package" for borderline personality disorder. The treatment package complies with the description agreed upon in common documents endorsed by all Danish Regions. The content of the treatment package includes psychotherapeutic treatment, according to the evidence based diagnose-specific manuals, and consultations with a psychiatrist. In this study this specifically includes, a treatment program consisting of dialectic behavioral treatment (DBT), delivered according to the manuals by Linehan, 1993 and Linehan, 2015.
  Interventions: Other: Treatment as usual
- The experimental intervention PEGASUS (Experimental): Patients in PEGASUS will, in addition to TAU, be offered to be affiliated with a case manager and to have their families involved in family-based interventions. Duration of the intervention will be nine months.
  The case manager will be a trained professional, who will be able to be a guiding figure and when needed, be able to help the patient contacting different authorities. The case manager can support the patient in solving everyday life problems, and will be an occupational therapist, a nurse, or a social worker. The case manager will offer the patients nine extra individual sessions during their treatment course.
  The format of the family-based interventions will be two psychoeducational workshops with 6 to 8 families invited and six multifamily group meetings, in which the patient and one or two relatives can participate. Theories behind Psychoeducational Multifamily Groups, Compassion Cultivation Training and Family Connections (FC, Hoffman et al., 2007) will be drawn upon.
  Interventions: Other: The experimental intervention PEGASUS

INTERVENTIONS:
Other: The experimental intervention PEGASUS — See arm description.
  Other Names: Case Manager; Family-based interventions
  Arms: The experimental intervention PEGASUS
Other: Treatment as usual — See arm description
  Arms: Treatment as usual (TAU)

SUMMARY:
The purpose of the PEGASUS study is to conduct a pilot trial to test the feasibility and acceptability of the PEGASUS intervention, adding a case manager and family-based interventions meetings to the existing psychiatric integrated care-models known as "Treatment Packages" in Denmark. We will conduct a randomized, assessor-blinded parallel-groups superiority clinical trial, testing the PEGASUS intervention for emotionally unstable personality disorder "EUPD", borderline type (borderline personality disorder) compared to "Treatment as Usual" before moving on to testing in a full-scale trial. Participants will be assessed at baseline and 9 month post baseline at study conclusion

DETAILED DESCRIPTION:
Background and rationale:

Unmet needs for patients diagnosed with emotionally unstable personality disorder (borderline personality disorder).

People with emotionally unstable personality disorder, borderline type, also known as borderline personality disorder (BPD) have substantial degrees of impairment (in educational, work, family, and social functioning) even after treatment, and they contribute very substantially to the burden of psychiatric disorders on a population level. When treatment in primary care is insufficient, these patients should be referred to psychiatric integrated care-models known as "treatment packages" in the secondary psychiatric healthcare sector. The treatment packages were introduced in Denmark in 2013. More than half of patients finishing a treatment package may still have symptoms, and it is also a clinical experience and hypothesis, that many patients will continue to receive more than one treatment package either for the same disorder or for different disorders. Furthermore, the level of functioning, particularly in BPD, often remains impaired despite symptomatic relief.

Family members are often both the first and the last line of defense, as they are the people whom the patient will contact 24/7, whenever there is an obstacle or a crisis related to the mental disorder. The lives of the family members are severely affected, as they may live in constant worry for their mentally ill relative, and they may need to be ready to throw everything else aside, when there is a crisis. Moreover, they will also often play the role as self-taught lawyers or case managers to help the patient to get the necessary treatment and to avoid severe social adversities.

Enhanced treatment, case management and involvement of families Over the last 25 years we have learned a great deal about the benefits of providing additional support for people with early psychosis. Our OPUS trial resulted in more than 40 publications, and has been highly cited (2700 citations, February 2023 (Web of Science)). We have learned from the OPUS trial, that prompt and skilled treatment for those with recent onset psychosis can improve health outcomes. The most important elements in the experimental OPUS-treatment were involvement of families and affiliation with a case manager. The results of the OPUS trial have been replicated in many countries, and there is now solid evidence for "Early Intervention Services", summarized in a meta-analysis and a recent Cochrane Review. A next obvious research question is, whether the same clinical approaches and treatment elements could be helpful for other mental health conditions. In a recent Australian study it was shown, that caregivers of young people with borderline personality features experience adversities similar to, or greater than, that reported by caregivers of young people with other severe illnesses. Currently, except from a single trial carried out with young people with BPD, and few trials investigating the effect of psychoeducation or group therapy with relatives, we lack an evidence base to know, if comparable comprehensive treatment packages can help the patients with BPD and their families.

Participants

We will recruit outpatients, who have been referred to the Psychotherapeutic Outpatient Department (POD), Mental Health Centre Glostrup, Mental Health Services of the Capital Region of Denmark. The patients must have been accepted in the treatment package for BPD. The patients will be able to bring 1-2 relatives to participate in the study.

Inclusion and written consent

Patients will be approached at their first meeting, after getting accepted into the treatment package program at POD. If interested, the patients will be scheduled for an inclusion meeting with a research assistant from the project, who is a trained physician. The inclusion meeting will take place uninterrupted in an office at the POD. Here participating patients will receive detailed written and oral information about participation, and give informed written consent.

In addition to this, the patient's relatives' experience of the PEGASUS intervention and TAU will be evaluated. The relatives' contact information will be obtained through the participating patients. They will be contacted by phone to schedule an inclusion meeting. The inclusion meeting will take place by phone call, where the relatives will receive detailed information about study participation and sign a digital version of the written consent.

The participants can withdraw their consent at any time during or after the study.

Assessment

We will be collecting data at inclusion to the study and at study conclusion after 9-month treatment. An additional follow up is under consideration, but not scheduled. Assessment will be conducted by semi structured interviews, questionnaires, collecting data from patient records and register based data from the Danish registers.

Calculation of sample size and analysis

In the main trial, we will have 90% power to detect a relevant difference of 7.2 (SD 19.2) on the WHODAS, which will require 2*150=300 participants with BPD. Based on this number of participants, it will be necessary to carry out a pilot trial with 15-20 participants in each arm. We will analyze all outcomes for safety and satisfaction. As per pilot trial guidelines, we will assess nominal differences regarding safety and acceptability. Safety will be defined through potential side effects, and whether the intervention group appears to get worse over time.

ELIGIBILITY:
Participating Patients

Inclusion Criteria:

* Must be able to give an informed written consent.
* Must be newly accepted in the pre-planned BPD treatment packages.
* ≥18 years of age.
* Agreeing to involvement of one or two informal caregivers, families, or close friends ("Relatives").
* Capable of reading and understanding Danish.

Exclusion Criteria:

* None*

  * Note that to get accepted into a treatment package for BPD, patients must not fulfill the criteria for a F20 diagnosis or the criteria for alcohol or substance abuse or harmful use.

Participating Relatives:

Inclusion Criteria:

* Must be able to give an informed written consent.
* ≥18 years of age.
* Capable of reading and understanding Danish.

Exclusion criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Level of functioning | Study inclusion and at 9 months at study completion
  WHODAS 2.0, 36-item interviewer-administered version (WHO's Disability Assessment Schedule). Measured in patients.

SECONDARY OUTCOMES:
Symptom relief | Study inclusion and at 9 months at study completion
  Measured by: Symptoms assessed with semi structured interviews using the Zanarini rating scale for borderline personality disorder (ZAN-BPD) and the personality disorder severity ICD-11 (PDS-ICD-11) and self-report by the borderline Symptom List 23 (BSL-23). Measured in patients.
Presences of suicidal ideations | Study inclusion and at 9 months at study completion
  Evaluated by the Suicidal Ideation Attributes Scale (SIDAS) and patient records. Measured in patients.
Well-being | Study inclusion and at 9 months at study completion
  Measured using WHO-5 (WHO-5 Questionnaires and Symptom Checklist 10 (SCL-10). Measured in patients and participating relatives.
Change in quality of relation between patient and relatives | Study inclusion and at 9 months at study completion
  Will be measured by using the Relationship Assessment scale General version (RAS-G). Measured in patients and participating relatives.
Ability to apply therapeutic tools learnt in therapy to everyday life situations. | At study inclusion and 9 months later at study conclusion
  The Dialectical Behavior Therapy Ways of Coping Checklist, Danish version (DBT-WCCL). Measured in patients and participating relatives.
Perceived burden by relatives | Study inclusion and at 9 months at study completion
  Evaluated by the relatives answering the Burden Assessment Scale (BAS). Measured only in relatives.
Satisfaction and acceptability of treatment | At study conclusion
  Measured with Client Satisfaction Questionnaire (CSQ)18, Process of Recovery Questionnaire (QPR)19 and Negative Effects questionnaire. As well as measuring treatment attendance and completion of the program. Measured in patients and participating relatives.
Patient Recorded Outcome Measures (PROM) | Study inclusion and at 9 months at study completion. Measured in patients
  Data from the local "Treatment Effect" database (Dansk: "Behandlingseffekt"). Including: Brief INSPIRE-O, Sheehan's Disability Scale (SDS), Level of Personality Functioning Scale Brief From 2.0 (LPFS BF 2.0).

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Hjorthøj, Ph.d., Principal Investigator — Copenhagen Research Center for Mental Health
Locations (1):
- Copenhagen Research Center for Mental Health - CORE, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Available upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After publication
Access Criteria: Upon request

REFERENCES:
- [Background] Leichsenring F, Heim N, Leweke F, Spitzer C, Steinert C, Kernberg OF. Borderline Personality Disorder: A Review. JAMA. 2023 Feb 28;329(8):670-679. doi: 10.1001/jama.2023.0589. PMID 36853245
- [Background] Hastrup LH, Kongerslev MT, Simonsen E. Low Vocational Outcome Among People Diagnosed With Borderline Personality Disorder During First Admission to Mental Health Services in Denmark: A Nationwide 9-Year Register-Based Study. J Pers Disord. 2019 Jun;33(3):326-340. doi: 10.1521/pedi_2018_32_344. Epub 2018 Mar 5. PMID 29505387
- [Background] Reinholt N, Hvenegaard M, Christensen AB, Eskildsen A, Hjorthoj C, Poulsen S, Arendt MB, Rosenberg NK, Gryesten JR, Aharoni RN, Alro AJ, Christensen CW, Arnfred SM. Transdiagnostic versus Diagnosis-Specific Group Cognitive Behavioral Therapy for Anxiety Disorders and Depression: A Randomized Controlled Trial. Psychother Psychosom. 2022;91(1):36-49. doi: 10.1159/000516380. Epub 2021 Jun 10. PMID 34111874
- [Background] McMain SF, Guimond T, Streiner DL, Cardish RJ, Links PS. Dialectical behavior therapy compared with general psychiatric management for borderline personality disorder: clinical outcomes and functioning over a 2-year follow-up. Am J Psychiatry. 2012 Jun;169(6):650-61. doi: 10.1176/appi.ajp.2012.11091416. PMID 22581157
- [Background] Muscroft J, Bowl R. The impact of depression on caregivers and other family members: Implications for professional support. http://dx.doi.org/101080/09515070050011105 2010; 13: 117-34.
- [Background] Senaratne R, Van Ameringen M, Mancini C, Patterson B. The burden of anxiety disorders on the family. J Nerv Ment Dis. 2010 Dec;198(12):876-80. doi: 10.1097/NMD.0b013e3181fe7450. PMID 21135638
- [Background] Lawn S, McMahon J. Experiences of family carers of people diagnosed with borderline personality disorder. J Psychiatr Ment Health Nurs. 2015 May;22(4):234-43. doi: 10.1111/jpm.12193. Epub 2015 Apr 8. PMID 25857849
- [Background] Petersen L, Jeppesen P, Thorup A, Abel MB, Ohlenschlaeger J, Christensen TO, Krarup G, Jorgensen P, Nordentoft M. A randomised multicentre trial of integrated versus standard treatment for patients with a first episode of psychotic illness. BMJ. 2005 Sep 17;331(7517):602. doi: 10.1136/bmj.38565.415000.E01. Epub 2005 Sep 2. PMID 16141449
- [Background] Correll CU, Galling B, Pawar A, Krivko A, Bonetto C, Ruggeri M, Craig TJ, Nordentoft M, Srihari VH, Guloksuz S, Hui CLM, Chen EYH, Valencia M, Juarez F, Robinson DG, Schooler NR, Brunette MF, Mueser KT, Rosenheck RA, Marcy P, Addington J, Estroff SE, Robinson J, Penn D, Severe JB, Kane JM. Comparison of Early Intervention Services vs Treatment as Usual for Early-Phase Psychosis: A Systematic Review, Meta-analysis, and Meta-regression. JAMA Psychiatry. 2018 Jun 1;75(6):555-565. doi: 10.1001/jamapsychiatry.2018.0623. PMID 29800949
- [Background] Puntis S, Minichino A, De Crescenzo F, Cipriani A, Lennox B, Harrison R. Specialised early intervention teams for recent-onset psychosis. Cochrane Database Syst Rev. 2020 Nov 2;11(11):CD013288. doi: 10.1002/14651858.CD013288.pub2. PMID 33135811
- [Background] Seigerman MR, Betts JK, Hulbert C, McKechnie B, Rayner VK, Jovev M, Cotton SM, McCutcheon L, McNab C, Burke E, Chanen AM. A study comparing the experiences of family and friends of young people with borderline personality disorder features with family and friends of young people with other serious illnesses and general population adults. Borderline Personal Disord Emot Dysregul. 2020 Jul 22;7:17. doi: 10.1186/s40479-020-00128-4. eCollection 2020. PMID 32704374
- [Background] Chanen AM, Betts JK, Jackson H, Cotton SM, Gleeson J, Davey CG, Thompson K, Perera S, Rayner V, Andrewes H, McCutcheon L. Effect of 3 Forms of Early Intervention for Young People With Borderline Personality Disorder: The MOBY Randomized Clinical Trial. JAMA Psychiatry. 2022 Feb 1;79(2):109-119. doi: 10.1001/jamapsychiatry.2021.3637. PMID 34910093
- [Background] Bateman A, Fonagy P. A randomized controlled trial of a mentalization-based intervention (MBT-FACTS) for families of people with borderline personality disorder. Personal Disord. 2019 Jan;10(1):70-79. doi: 10.1037/per0000298. Epub 2018 Jul 12. PMID 29999394
- [Background] Pearce J, Jovev M, Hulbert C, McKechnie B, McCutcheon L, Betts J, Chanen AM. Evaluation of a psychoeducational group intervention for family and friends of youth with borderline personality disorder. Borderline Personal Disord Emot Dysregul. 2017 Mar 24;4:5. doi: 10.1186/s40479-017-0056-6. eCollection 2017. PMID 28352470
- [Background] Grenyer BFS, Bailey RC, Lewis KL, Matthias M, Garretty T, Bickerton A. A Randomized Controlled Trial of Group Psychoeducation for Carers of Persons With Borderline Personality Disorder. J Pers Disord. 2019 Apr;33(2):214-228. doi: 10.1521/pedi_2018_32_340. Epub 2018 Mar 5. PMID 29505385
- [Background] Flynn D, Kells M, Joyce M, Corcoran P, Herley S, Suarez C, Cotter P, Hurley J, Weihrauch M, Groeger J. Family Connections versus optimised treatment-as-usual for family members of individuals with borderline personality disorder: non-randomised controlled study. Borderline Personal Disord Emot Dysregul. 2017 Aug 30;4:18. doi: 10.1186/s40479-017-0069-1. eCollection 2017. PMID 28861273
- [Background] Bohus M, Kleindienst N, Limberger MF, Stieglitz RD, Domsalla M, Chapman AL, Steil R, Philipsen A, Wolf M. The short version of the Borderline Symptom List (BSL-23): development and initial data on psychometric properties. Psychopathology. 2009;42(1):32-9. doi: 10.1159/000173701. Epub 2008 Nov 20. PMID 19023232
- [Background] Linehan MM. Skills training manual for treating borderline personality disorder. New York: Guilford Press, 1993.
- [Background] Linehan M. DBT skills training manual, Second edition. New York: The Guilford Press, 2015.
- [Background] McFarlane WR, Lukens E, Link B, Dushay R, Deakins SA, Newmark M, Dunne EJ, Horen B, Toran J. Multiple-family groups and psychoeducation in the treatment of schizophrenia. Arch Gen Psychiatry. 1995 Aug;52(8):679-87. doi: 10.1001/archpsyc.1995.03950200069016. PMID 7632121
- [Background] Hansen NH, Juul L, Pallesen KJ, Fjorback LO. Effect of a Compassion Cultivation Training Program for Caregivers of People With Mental Illness in Denmark: A Randomized Clinical Trial. JAMA Netw Open. 2021 Mar 1;4(3):e211020. doi: 10.1001/jamanetworkopen.2021.1020. PMID 33683334
- [Background] https://www.regioner.dk/media/5559/pakkeforloeb-for-emotionel-ustabil-personlighedsforstyrrelse.pdf